CLINICAL TRIAL: NCT00145288
Title: Prospective Study of Patients Med Hirsutism as Primary Work Diagnose
Brief Title: Prospective Study of Patients With Hirsutism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: 010
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Hirsutism; Type 2 Diabetes; Polycystic Ovary Syndrome
Keywords: hirsutism; type 2 diabetes; polycystic ovary syndrome; metabolism
MeSH Terms: conditions — Hirsutism; Diabetes Mellitus, Type 2; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hirsutism is the presence of terminal hairs in a male-like pattern in females, due to elevated male hormone levels. Females with hirsutism are often overweight and have metabolism disturbances as insulin resistance and impaired glucose tolerance.

The previous studies showed that patients with hirsutism (especially them with polycystic ovarian syndrome (PCOS)) have an increased risk to develop type 2 diabetes mellitus on the background of insulin resistance / hyperinsulinemia: 30-35 % of females with PCOS had impaired glucose tolerance and 5-10 % of them diabetes. Hyperinsulinemia increases the risk to develop dyslipidemia and cardiovascular diseases.

A previous study in our department who included 340 females with hirsutism (210 with idiopathic hirsutism and 134 with PCOS) showed that 6.6% of them had diabetes and 55% insulin resistance.

There were only few long-term follow up studies of patients with hirsutism concerning their risk to develop diabetes. As far as we now, such studies on patients with idiopathic hirsutism are not available until now.

Hirsutism is been treated with low dose oral contraceptives, which are suppressing androgen production. This treatment can also influence the risk to develop diabetes and atheromatosis. The previous studies showed that the low dose oral contraceptives had modest influence on the lipid profiles and carbohydrate metabolism in patients with hirsutism, but increased the risk to develop coronary disease.

Aim

* To study and quantify, in patients with hirsutime, the risk to develop type 2 diabetes on the background of insulin resistance / decreased glucose tolerance and atheromatosis on the background of insulin resistance / hypercholesterolemia.
* To clarify the effect of P-pills on patients hair growth and metabolism.

DETAILED DESCRIPTION:
Hirsutism is the presence of terminal hairs in a male-like pattern in females, due to elevated male hormone levels. Females with hirsutism are often overweight and have metabolism disturbances as insulin resistance and impaired glucose tolerance.

The previous studies showed that patients with hirsutism (especially them with polycystic ovarian syndrome (PCOS)) have an increased risk to develop type 2 diabetes mellitus on the background of insulin resistance / hyperinsulinemia: 30-35 % of females with PCOS had impaired glucose tolerance and 5-10 % of them diabetes (1, 2, 3, 4). Hyperinsulinemia increases the risk to develop dyslipidemia and cardiovascular diseases (5, 6, 7, 8, 9).

A previous study in our department who included 340 females with hirsutism (210 with idiopathic hirsutism and 134 with PCOS) showed that 6.6% of them had diabetes and 55% insulin resistance (10).

There were only few long-term follow up studies of patients with hirsutism concerning their risk to develop diabetes. As far as we now, such studies on patients with idiopathic hirsutism are not available until now.

Hirsutism is been treated with low dose oral contraceptives, which are suppressing androgen production. This treatment can also influence the risk to develop diabetes and atheromatosis. The previous studies showed that the low dose oral contraceptives had modest influence on the lipid profiles and carbohydrate metabolism in patients with hirsutism, but increased the risk to develop coronary disease (11).

Aim

* To study and quantify, in patients with hirsutime, the risk to develop type 2 diabetes on the background of insulin resistance / decreased glucose tolerance and atheromatosis on the background of insulin resistance / hypercholesterolemia.
* To clarify the effect of P-pills on patients hair growth and metabolism.

Design The patients who had previously included in the study between1997 - 2000 (231) will be contacted in order to be followed. We will estimate the grad of excess hair growth, the hormonal and metabolism profiles.

Inclusion criteria The patients which had been included in the previous study between 1997 - 2000, oral glucose tolerance test included.

Exclusion criteria Pregnancy.

Investigations

Anamnesis: previous treatment, pregnancy / in-utero fertilisation history, family predisposition to diabetes and cardiovascular diseases.

Clinical examination: Ferriman-Gallwey score, body mass index (BMI), waist / hip ratio (WHR), blood pressure.

Blood analyses:

* Metabolism profile (oral glucose tolerance test, lipid profile);
* Hormonal profile (androgen and oestrogen levels, prolactin, FH, FSH).

The ethic aspects

We want to evaluate the effect of the treatment and how the risk factors are influenced by the treatment.

All the patients will receive both oral and written information about the study. It will be emphasised at participation is voluntary and the informed consent can be retracted at any time and this will not influence the treatment of them.The trial is validated by the local ethics committee.

The project will be carried on The Endocrinology Department, Odense University Hospital, Denmark, which will supply technical assistance. Blood analyses will be founded by private founds.

References

1. Diamanti-Kandarakis, E., Baillargeon, J. P., Iuorno, M. J., Jakubowicz, D. J., and Nestler, J. E. A modern medical quandary: polycystic ovary syndrome, insulin resistance, and oral contraceptive pills.J.Clin.Endocrinol.Metab 2003 88 1927-1932
2. Arslanian, S. A., Lewy, V. D., and Danadian, K. Glucose intolerance in obese adolescents with polycystic ovary syndrome: roles of insulin resistance and beta-cell dysfunction and risk of cardiovascular disease.J.Clin.Endocrinol.Metab 2001 86 66-71
3. Ehrmann, D. A., Barnes, R. B., Rosenfield, R. L., Cavaghan, M. K., and Imperial, J. Prevalence of impaired glucose tolerance and diabetes in women with polycystic ovary syndrome.Diabetes Care 1999 22 141-146
4. Palmert, M. R., Gordon, C. M., Kartashov, A. I., Legro, R. S., Emans, S. J., and Dunaif, A. Screening for abnormal glucose tolerance in adolescents with polycystic ovary syndrome.J.Clin.Endocrinol.Metab 2002 87 1017-1023
5. Elting, M. W., Korsen, T. J., Bezemer, P. D., and Schoemaker, J. Prevalence of diabetes mellitus, hypertension and cardiac complaints in a follow-up study of a Dutch PCOS population.Hum.Reprod. 2001 16 556-560
6. Loucks, T. L., Talbott, E. O., McHugh, K. P., Keelan, M., Berga, S. L., and Guzick, D. S. Do polycystic-appearing ovaries affect the risk of cardiovascular disease among women with polycystic ovary syndrome?Fertil.Steril. 2000 74 547-552
7. Mather, K. J., Kwan, F., and Corenblum, B. Hyperinsulinemia in polycystic ovary syndrome correlates with increased cardiovascular risk independent of obesity.Fertil.Steril. 2000 73 150-156
8. Vrbikova, J., Cifkova, R., Jirkovska, A., Lanska, V., Platilova, H., Zamrazil, V., and Starka, L. Cardiovascular risk factors in young Czech females with polycystic ovary syndrome.Hum.Reprod. 2003 18 980-984
9. Wild, S., Pierpoint, T., McKeigue, P., and Jacobs, H. Cardiovascular disease in women with polycystic ovary syndrome at long-term follow-up: a retrospective cohort study.Clin.Endocrinol.(Oxf) 2000 52 595-600
10. Glintborg, D., Henriksen, J. E., Andersen, M., Hagen, C., Hangaard, J., Rasmussen, P. E., Schousboe, K., and Hermann, A. P. Prevalence of endocrine diseases and abnormal glucose tolerance tests in 340 Caucasian premenopausal women with hirsutism as the referral diagnosis.Fertil.Steril. 2004 82 1570-1579
11. Creatsas, G., Koliopoulos, C., and Mastorakos, G. Combined oral contraceptive treatment of adolescent girls with polycystic ovary syndrome. Lipid profile.Ann.N.Y.Acad.Sci. 2000 900 245-252

ELIGIBILITY:
Inclusion Criteria:

* The patients which had been included in the previous study between 1997 - 2000, oral glucose tolerance test included.

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340
Dates: Start 2003-10; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Andries, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark